CLINICAL TRIAL: NCT04032574
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Parallel Group Trial to Evaluate the Efficacy and Tolerability of a Phytotherapy Combination (Aqualibra) in Patients With Uncomplicated Cystitis
Brief Title: Efficacy and Tolerability of a Phytotherapy Combination (Aqualibra) in Patients With Uncomplicated Cystitis
Acronym: AquUTI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medice Arzneimittel Pütter GmbH & Co KG (Industry)
Collaborators: Dr. Wiedey GmbH - Institut Für Klinische Forschung (Unknown); Medidata Dr. Möller GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 97.019/91
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Urinary Tract Infection Lower Acute

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Herbal medicinal product (Experimental): three times daily two film coated tablets containing: extracts of restharrow root (Ononidis radix) 80mg,Java tea (Orthosiphonis folium) 90mg, goldenrod herb (Solidaginis herba) 180mg
  Interventions: Combination Product: Herbal Medicinal Product
- Placebo (Placebo Comparator): three times daily two film coated tablets
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: Herbal Medicinal Product
  Arms: Herbal medicinal product
Other: Placebo
  Arms: Placebo

SUMMARY:
This randomized, placebo-controlled, double-blind study investigated the efficacy and safety of the herbal medicinal product containing a combination of extracts of restharrow root (Ononidis radix), Java tea (Orthosiphonis folium) and goldenrod herb (Solidaginis herba) in women with acute lower uUTI.

DETAILED DESCRIPTION:
This randomized, placebo-controlled, double-blind study investigated the efficacy and safety of the herbal medicinal product containing a combination of extracts of restharrow root (Ononidis radix), Java tea (Orthosiphonis folium) and goldenrod herb (Solidaginis herba) in the treatment of acute lower uUTI. The herbal medicinal product represent a multi-target therapy that includes diuretic, anti-inflammatory and antimicrobial aspects.

Patients were randomized to one of the two treatment groups and treated with the phytotherapeutic agent or matching placebo for seven days.

The primary endpoint was microbiologic response defined as reduction in bacterial urine culture counts by at least 10*2 CFU/ml.

ELIGIBILITY:
Inclusion Criteria:

* Female outpatients aged 18-75 years
* Diagnosis of acute lower uUTI occurring for the first time or acute relapse of chronic recurrent uUTI
* Typical symptoms of cystitis (pollakisuria, dysuria and urgency)
* Bacterial count of 10*4 - 10*6 colony forming units (CFU)/mL in midstream urine
* Presence of >20 leukocytes/µL of urine measured by dipstick test
* No antibiotic treatment required according to the investigator
* Women of childbearing potential were allowed to participate only if they used a highly effective method of contraception
* Written informed consent

Exclusion Criteria:

* Known hypersensitivity to any of the active substances or excipients of the study medication
* Antibiotic treatment during the past 8 days or indication for antibiotic treatment for the current infection
* Patients with trichomoniasis, chlamydiosis or gonorrhoea
* Use of concomitant medication that may have an effect on the UTI, including other phytotherapeutics with similar effects, saluretics (including those in antihypertensives) or other drugs with a similar mode of action, urinary acidifying agents (e.g. Acimethin®), antibiotics, or phytotherapeutics with possible antibiotic effects
* Patients with suspected ovarian inflammation (e.g. adnexitis)
* Patients with suspected renal inflammation (e.g. pyelonephritis)
* Patients with complicated UTI (e.g. obstruction, stones, reflux)
* Patients with overactive bladder
* Patients with vegetative urogenital syndrome
* Patients who were currently participating or had participated in another clinical trial within 30 days before enrolment
* Patients in poor general condition
* Alcohol- or drug-addicted patients
* Pregnant or nursing women or women not using highly effective methods of contraception
* Patients with mental illness or no/limited legal capacity
* Patients held in an institution by legal or official order
* Patients who were not proficient in spoken or written German
* Patients with a urine bacterial count >10*6 CFU/mL were to be excluded from further participation in the study unless they specifically wished to continue treatment with the study medication.
* No contraindications against the study medication were known at the time of study protocol preparation

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 1991-10-08 (Actual); Primary Completion 1992-03-27 (Actual); Study Completion 1992-03-27 (Actual)

PRIMARY OUTCOMES:
microbiologic response | 7 days
  Percentage of patients with a reduction in bacterial urine culture counts by at least 10*2 CFU/ml

SECONDARY OUTCOMES:
Leukocyturia | 7 days
  Percentage of patients without leukocyturia

CONTACTS AND LOCATIONS:
Overall Officials: Roland Fischer, PhD, Study Director — Medice Arzneimittel Pütter GmbH & CoKG

REFERENCES:
- [Derived] Vahlensieck W, Lorenz H, Schumacher-Stimpfl A, Fischer R, Naber KG. Effect of a Herbal Therapy on Clinical Symptoms of Acute Lower Uncomplicated Urinary Tract Infections in Women: Secondary Analysis from a Randomized Controlled Trial. Antibiotics (Basel). 2019 Dec 7;8(4):256. doi: 10.3390/antibiotics8040256. PMID 31817885